CLINICAL TRIAL: NCT06757933
Title: Comparison Of Spencer Technique And Isotonic Exercise In Patients With Adhesive Capsulitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/771
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Adhesive Capsulitis, Shoulder
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group I (Experimental)
  Interventions: Combination Product: The Spencer technique
- Interventional group II (Experimental)
  Interventions: Combination Product: isotonic workouts

INTERVENTIONS:
Combination Product: The Spencer technique — The Spencer technique, which consists of seven different manual movements intended to increase shoulder mobility and lessen pain, was used to treat the participants in this group. The method seeks to improve blood flow, loosen up the shoulder joint and soft tissues, and reduce any tightness or impingement that is causing pain in the sub-acromial area. By re-establishing appropriate shoulder function and movement patterns, the Spencer approach is commonly used to treat disorders including adhesive capsulitis.
  Arms: Interventional group I
Combination Product: isotonic workouts — This group's members engaged in isotonic workouts that emphasized forward flexion and extension motions. Both concentric (shortening the muscle) and eccentric (lengthening the muscle) motions were used in these exercises. These exercises were designed to increase shoulder range of motion and strengthen the rotator cuff muscles. People with Adhesive Capsulitis may have less pain and have better shoulder function if they perform isotonic workouts, which increase muscular strength and stability.
  Arms: Interventional group II

SUMMARY:
This study examines the efficacy of two forms of therapy for Adhesive Capsulitis, a condition characterized by stiffness, pain, and limited mobility in the shoulder joint. It is also commonly known as "Frozen Shoulder".

DETAILED DESCRIPTION:
Patients between the ages of 30 and 55 were randomly assigned to one of two groups for the trial held at the Saleem Free Hospital Okara and Dar-ul-Shifa Hospital. Group 2 engaged in isotonic exercises that emphasized concentric and eccentric motions of forward flexion and extension, whereas Group 1 was given the Spencer approach, which involved seven different movements. A goniometer and the Numeric Pain Rating Scale were used to measure the range of motion and pain. SPSS 20 was used to analyze the data and assess how well the treatments worked. The findings provided light on how well manual therapy and exercise compare in terms of reducing pain and increasing shoulder movement in people with adhesive capsulitis.

ELIGIBILITY:
Inclusion Criteria

* Both genders aged 30-55 years
* Unilateral Adhesive Capsulitis
* Pain lasting for more than one month
* Capsular pattern of motion restriction
* Diabetic patients were included.

Exclusion Criteria

* Participants with rotator cuff tear
* Rheumatoid and gouty arthritis
* Tumors of the shoulder region
* Peripheral nerve injuries
* Shoulder girdle fracture and dislocation
* History of shoulder surgery were excluded.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2025-03-02 (Estimated)

PRIMARY OUTCOMES:
The Numeric Pain Rating Scale | 12 Months
  (NPRS) was used to measure the subjects' level of pain. This scale helps measure the amount of pain alleviation attained with each intervention by allowing participants to rank their discomfort from 0 (no pain) to 10 (worst possible pain).
goniometer | 12 Months
  A goniometer, which measures the angle of joint movement, was used to measure the shoulder's range of motion (ROM). Improvements in shoulder mobility, which is frequently limited in adhesive capsulitis, were assessed with the aid of this assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Saleem Memorial Free Hospital Address: College road, Depalpur Rd, adjacent baldia hall, Okara, Okāra, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No